CLINICAL TRIAL: NCT03031158
Title: Pilot Trial of a Hip-spine Intervention for Older Adults With a Primary Complaint of Low Back Pain
Brief Title: Hip-spine Intervention for Older Adults With Chronic Low Back Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Gregory Evan Hicks, Associate Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 943328
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SFEX+H (Experimental): Participants will receive an intervention consisting of heat to the low back, manual therapy to the hip (including movement of the hip by the therapist), hip-focused strengthening exercises and a trunk muscle training program including exercises for the abdominal and low back muscles.
  Interventions: Behavioral: SFEX+H
- SFEX (Active Comparator): Participants will receive an intervention consisting of heat to the low back, manual therapy to the hip (including movement of the hip by the therapist) and a trunk muscle training program including exercises for the abdominal and low back muscles.
  Interventions: Behavioral: SFEX

INTERVENTIONS:
Behavioral: SFEX+H — Participants will receive an intervention consisting of heat to the low back, manual therapy to the hip (including movement of the hip by the therapist), hip-focused strengthening exercises and a trunk muscle training program including exercises for the abdominal and low back muscles. The intervention will be delivered twice weekly for 8 weeks.
  Arms: SFEX+H
Behavioral: SFEX — Participants will receive an intervention consisting of heat to the low back, manual therapy to the hip (including movement of the hip by the therapist) and a trunk muscle training program including exercises for the abdominal and low back muscles. The intervention will be delivered twice weekly for 8 weeks.
  Arms: SFEX

SUMMARY:
Low back pain (LBP) is extremely common in older adults and is associated with a host of negative consequences, including decreased physical function and increased healthcare utilization. Among older adults with LBP, hip impairments indicative of hip joint disease are more prevalent and associated with greater disability than among older adults without LBP. This study will investigate a novel intervention designed to improve LBP-related disability by combining a typical spine-focused exercise program with a hip-focused intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age 60-85
2. Low Back Pain for ≥ 3 months with pain of at least moderate intensity every day or almost every day that requires activity modification.
3. Presence of at least 1 hip impairment denoted by the American College of Rheumatology as potential indicators of hip osteoarthritis: hip pain, pain on hip internal rotation or morning stiffness of the hip of <60 minutes.

Exclusion Criteria:

1. Previous hip fracture repair or total hip replacement
2. Prominent component of radicular pain: CLBP with distal radiation below the knee
3. Known spinal pathology other than osteoarthritis: (e.g., a history of back surgery or recent trauma, spinal stenosis, vertebral compression fractures, ankylosing spondylitis, carcinoma metastatic to the spine)
4. Non-ambulatory, or severely impaired mobility (i.e., require the use of a wheelchair)
5. Folstein Mini-Mental State Examination score of <24
6. Severe visual or hearing impairment.
7. Red flags indicative of a serious disorder underlying the LBP: Red flags that would require specialized medical attention include fever, significant unintentional weight loss, a sudden recent change in the character or intensity of pain, trauma that preceded the onset of pain, or signs and symptoms of caudae equinae (i.e. loss of sensation over saddle region, significant disturbances in bowel and bladder function).
8. Significant pain in parts of the body other than the back or acute LBP.
9. Acute, ongoing illness.
10. Inability to participate in the study for the full six months for any known reason.(i.e. moving away, extended vacation)
11. Received physical therapy for their LBP within in the last 3 months.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-03-13 (Actual); Study Completion 2018-03-13 (Actual)

PRIMARY OUTCOMES:
Quebec Low Back Pain Disability Scale | Change in disability score from pre-intervention to 20 weeks later
Patient-Specific Functional Scale | Change in pain-related function score from pre-intervention to 20 weeks later

SECONDARY OUTCOMES:
Walking Endurance as measured by the 6 minute walk test | Change in walking endurance from pre-intervention to 20 weeks later
Walking speed | Change in walking endurance from pre-intervention to 20 weeks later

CONTACTS AND LOCATIONS:
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No